CLINICAL TRIAL: NCT01116141
Title: A Phase II, Multi-center, Randomized, Parallel Group, Double-blind, MTX Controlled Study to Assess the Clinical Efficacy, Safety and Tolerability of CH-4051 in Patients With Active RA Who Have Shown an Inadequate Response to MTX Monotherapy
Brief Title: A Study of CH-4051 in Patients With Rheumatoid Arthritis (RA)
Acronym: MOTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chelsea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CH-4051-RA202
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; MTX; CH-405; antifolates
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Methotrexate (MTX) + Folic Acid (Active Comparator): 20 mg MTX weekly + 1 mg folic acid daily
  Interventions: Drug: Methotrexate (MTX); Drug: Folic Acid
- 0.3 mg CH-4051 (Experimental): 0.3 mg CH-4051 daily
  Interventions: Drug: CH-4051
- 1.0 mg CH-4051 (Experimental): 1.0 mg CH-4051 daily
  Interventions: Drug: CH-4051
- 3.0 mg CH-4051 (Experimental): 3.0 mg CH-4051 daily
  Interventions: Drug: CH-4051
- 3.0 mg CH-4051 + folic acid (Experimental): 3.0 mg CH-4051 + 1.0 mg folic acid daily
  Interventions: Drug: CH-4051; Drug: Folic Acid

INTERVENTIONS:
Drug: CH-4051 — Different doses CH-4051 to be compared
  Arms: 0.3 mg CH-4051; 1.0 mg CH-4051; 3.0 mg CH-4051; 3.0 mg CH-4051 + folic acid
Drug: Methotrexate (MTX) — 20 mg MTX weekly
  Other Names: amethopterin
  Arms: Methotrexate (MTX) + Folic Acid
Drug: Folic Acid — 1 mg folic acid daily
  Other Names: folate
  Arms: 3.0 mg CH-4051 + folic acid; Methotrexate (MTX) + Folic Acid

SUMMARY:
The purpose of this study is to determine if CH-4051 is a safe and effective treatment for rheumatoid arthritis.

DETAILED DESCRIPTION:
Multi-center, multi-national, double-blind, randomized, active-controlled (MTX), 3-month study with 4 doses of CH-4051 (0.3 mg, 1.0 mg, 3.0 mg and 3.0 mg with 1mg of folic acid supplementation p.o. daily) compared to a "standard" dose of MTX at 20 mg per week with 1 mg of folic acid supplementation p.o. daily. This study will be conducted in two parts:

Part A: Patients will be randomized to 0.3 mg CH-4051, 1.0 mg CH-4051 or MTX. Part B: Patients will not be randomized into Part B until the Data Monitoring Committee has reviewed safety data from the Part A when approximately 25 patients (10 patients in each CH-4051 dose groups and 5 patients in the MTX groups) have completed 3 months of treatment. At this time the DMC will make a recommendation whether or not to commence randomization to 3.0 mg CH-4051, 3.0 mg CH-4051 with 1.0 mg of folic acid.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between the ages of 18 and 80;
* Have diagnosed active rheumatoid arthritis according to ACR criteria functional class I-III;
* Have at least 6 swollen joints (max = 66) and 6 tender joints (max = 68) at screening and baseline visits;
* Patients must have at least one of the following:
* C-reactive protein > 1.0 mg/dl at screening;
* erythrocyte sedimentation rate > 28 mm/Hr;
* Patients must have been taking methotrexate between 15 and 25 mg/week for at least 3 months and at a stable dose for at least 6 weeks;
* Patients must be either Rheumatoid Factor (RF) or anti-cyclic citrullinated peptide (anti-CCP) positive;
* Patients must have voluntarily signed the informed consent.

Exclusion Criteria:

* Patients who received previous therapy with any biologic agent;
* Patients currently taking any disease modifying anti-rheumatic drug (DMARD) other than MTX;
* Previous non-biologic DMARD therapy is permitted as long as their last dose was at least 30 days prior to baseline;
* Female patients of child bearing potential who are pregnant or who are not using two methods of contraception (at least one barrier: i.e. condom) with their partner;
* Male patients who are sexually active and not using two methods of contraception (at least one barrier: i.e. condom) with their partner;
* Patients with any current active infection or infections requiring IV drug therapy within 30 days of baseline or oral therapy within 15 days of Baseline;
* Patients that have had any surgical procedures within 30 days of baseline;
* Patients with a history of HIV;
* Patients with Hepatitis B surface antigen positive and/or Hepatitis C antibody positive;
* Patients who consume more than 4 units of alcohol per week (1 unit = 5 ounces/150 ml of wine = 1.5 ounces/45 ml spirits = 12 ounces/360 ml of beer);
* Patients currently receiving any investigational drug or have received an investigational drug within 30 days of baseline or 5 half-lives of the investigational drug (whichever is longer);
* Patients with a history of cancer within the past 5 years other than a successfully treated, non-metastatic cutaneous squamous cell or basal cell carcinoma or cervical cancer in situ;
* Patients with a history of, or any, disease associated with an inflammatory arthritis other than RA;
* Patients with pulmonary fibrosis (Chest x-ray must be taken within 28 days of screening);
* Patients receiving probenecid;
* Patients who have received any steroid injections within 30 days of baseline;
* Patients with concomitant diseases that are unstable (i.e. cardiac, pulmonary) or that may affect drug activity (i.e. absorption, reactions, change in kinetics);
* Patients, in the investigator's opinion, that have any significant renal or hepatic impairment;
* Patients with a serum creatinine level > 1.5 mg/dl at screening;
* Patients with an ALT >1.5 ULN at screening;
* Patients considered by the investigator to be an unsuitable candidate to receive CH-4051;
* Wheelchair or bed-bound patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Co-primary: Hybrid American College of Rheumatology response criteria (hACR)followed by the ACR20 | 12 weeks
  The hybrid ACR (hACR) response was developed by the American College of Rheumatology to provide an improvement measure more sensitive to change than many other currently used measures, e.g., traditional ACR 20, 50 and 70 responses, while still maintaining clinical meaning. While traditional ACR 20, 50 and 70 response criteria are dichotomous measures (responder = yes/no), the hACR is a semi-continuous variable based upon the traditional ACR response but incorporating additional information on patient response into the outcome measure.

SECONDARY OUTCOMES:
DAS28 | 12 weeks
  The disease activity score (DAS) is a combined index that was developed in Nijmegen in the 1980s to measure the disease activity in patients with RA. It has been extensively validated for its use in clinical trials in combination with the European League Against Rheumatism (EULAR) response criteria.
ACR response criteria | 12 weeks
  ACR assessment criteria is a widely accepted composite index of improvement in RA proposed by the American College of Rheumatology (ACR). ACR20 refers to a composite improvement of 20% in swollen joint count, tender joint count, and 3 or more of the following 5 measures: patient's own global assessment of RA disease activity; physician's global assessment of disease activity; patient's own assessment of pain due to RA; acute-phase reactant (erythrocyte sedimentation rate (ESR) or CRP); and patient's self-assessed disability (Health Assessment Questionnaire).
Morning stiffness | 12 weeks
  Morning stiffness is a common complaint of patients suffering from rheumatoid arthritis. Severity and joints involves varies from patient to patient. Patients will be asked, "Over the past 7 days, what has been the duration of stiffness of your joints in the morning?" The amount of time it takes a patient's morning stiffness to subside will be captured in hours and minutes.
Safety and tolerability of CH-4051 in RA patients as determined by the frequency and severity of adverse events, laboratory abnormalities, and dropouts due to AEs | 12 weeks
  Safety will be assessed by physical exams, vital signs, laboratory safety (blood and urine) and AEs. Liver functions tests will be identified as laboratory values of particular interest.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur A Kavanaugh, MD, Principal Investigator